CLINICAL TRIAL: NCT06998173
Title: Phase 1 Study to Evaluate the Safety, Tolerability and Pharmacokinetics of DAT-1604 Tablets as Monotherapy in the Advanced Solid Tumor
Brief Title: Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of DAT-1604 in Advanced Solid Tumor
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Danatlas Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Danatlas Pharmaceuticals
Record Dates: First submitted 2025-05-16; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumors
Keywords: Polθ Inhibitor; Advanced Solid Tumors; Metastatic Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1, Dose escalation (Experimental): The part 1 is the dose escalation study, and set 6 dose level cohorts.On day 1 of cycle 1(C0D1), The patient takes DAT-1645 orally one time (single use) at the dose level in his or her enrollment cohort . Since C1D1(C0D4)，the DAT-1604 tablet is administered orally once daily at same dose level for 21 days per treatment cycle. Treatment continues until disease progression, or toxicity intolerance, or withdrawal from the study, or loss to follow-up, or initiation of new antitumor therapy, whichever occurs first.
  Interventions: Drug: DAT-1604 tablet
- Module 1 Part 2, dose expansion study to assess the food effects on pharmacokinetics（PK）. (Experimental): On day 1 of cycle 0 (C0D1), a single recommended oral dose of DAT-1604 is administered in the fasted state, withing a drug-free washout period of day 2 and day 3, and a single same dose of DAT-1604 is administered in the postprandial state on C0D4, with elution of the drug by C0D5, C0D6. Since C1D1(C0D7) , the DAT-1604 is administered orally once daily at the same dosage level, for 21 days as 1 treatment cycle , administered until disease progression, or toxicity intolerance, or withdrawal from the study, or loss to follow-up, or initiation of new antitumor therapy, or trial closure/termination, whichever occurs first.
  Interventions: Drug: DAT-1604 tablet
- Module 2 Part 2, optimized dose expansion (Experimental): The study sets two recommended dose levels. The patient will receive one of the dose levels, and be administered orally once daily at the same dosage level, for 21 days as 1 treatment cycle , administered until disease progression, or toxicity intolerance, or withdrawal from the study, or loss to follow-up, or initiation of new antitumor therapy, or trial closure/termination, whichever occurs first.
  Interventions: Drug: DAT-1604 tablet
- Module 3 Part 2, RP2D expansion (Experimental): The patient will be administered DAT-1604 with recommended phase 2 dose (RP2D) level, orally once daily , for 21 days as 1 treatment cycle , and administered until disease progression, or toxicity intolerance, or withdrawal from the study, or loss to follow-up, or initiation of new antitumor therapy, or trial closure/termination, whichever occurs first.
  Interventions: Drug: DAT-1604 tablet

INTERVENTIONS:
Drug: DAT-1604 tablet — DAT-1604, a potent and selective oral small molecule inhibitor of DNA Polymerase θ (Pol θ).

SUMMARY:
The primary objective of the study is to evaluate the safety, tolerability, PK, and preliminary efficacy of a Polθ Inhibitor DAT-1604 in patients with advanced/metastatic solid tumors, which is refractory to standard therapies, or for which no standard therapies exist.

DETAILED DESCRIPTION:
In Part 1, 6 dose cohorts will be set and defined maximum tolerated dose(MTD)/recommended dose for expansion (RDE). In Part 2, Food effects on pharmacokinetic of DAT-1604 will be assessed at RDE, and dose optimization will be conducted to definite recommended phase 2 dose (RP2D). Then , The RP2D expansion will be conducted in another 3 cohorts to evaluate the efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Male or female aged ≥18 years.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1.
4. Advanced or metastatic solid tumor, which is refractory to standard therapies, or for which no standard therapies exist.
5. Non-irradiated tumor tissue sample (archival or newly obtained core biopsy of a tumor lesion) available for submission for analysis.
6. Discontinued all previous treatments for cancer for at least 21 days or 5 half-lives, whichever is shorter, and recovered from the acute effects of therapy. Palliative radiotherapy must have completed 1 week prior to start of study treatment.
7. At least 1 radiologically evaluable lesion (measurable and/or non-measurable) that can be assessed at baseline and is suitable for repeated radiological evaluation by RECIST v1.1 for subjects.
8. Acceptable hematologic, renal, hepatic, and coagulation functions independent of transfusions and granulocyte colony-stimulating factor indicated by the following laboratory values:

   * Hemoglobin (Hgb) greater than or equal to 10 g/dL;
   * Leukocytes greater than or equal to 3,000/mcL;
   * Absolute neutrophil count greater than or equal to 1,500/mcL;
   * Platelets greater than or equal to 100,000/mcL;
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2 × upper limit of normal (ULN); if liver metastases, then ≤ 3 × ULN;
   * Bilirubin ≤ 1.5 × ULN; < 2 × ULN if hyperbilirubinemia is due to Gilbert's syndrome;
   * Serum albumin ≥ 30 g/L (3.0 g/dL);
   * Creatinine clearance ≥ 60 mL/min (Cockcroft-Gault Equation).
9. Willingness to abide by protocol defined contraceptive requirements for the duration of the study.
10. Estimated life expectancy of ≥12 weeks.

    -

Exclusion Criteria:

1. Subjects who are pregnant.
2. Subjects with Myelodysplastic syndrome (MDS)/Acute myeloid leukemia (AML) or with features suggestive of MDS/AML.
3. Have ongoing interstitial lung disease or pneumonitis.
4. Have any major gastrointestinal issues that could impact absorption of DAT-1604.
5. Subjects with brain metastases (subjects with treated brain metastases could be eligible if follow-up brain imaging after central nervous system-directed therapy shows no evidence of progression at least more than 4 weeks without neuropsychiatric symptom).
6. Have received a live vaccine within 30 days before the first dose of study treatment.
7. Recent major surgery within 4 weeks prior to entry into the study.
8. Have a history of allergy or hypersensitivity to study drug components.
9. Persistent toxicities ([CTCAE] Grade > 1) from prior anticancer therapy, excluding alopecia and CTCAE Grade 2 peripheral neuropathy.
10. Any of the following ECG findings at Screening, Admission and/or pre dose on Day 1:

    * Any out of range ECG parameter(s) or abnormal finding(s) considered clinically significant by the Investigator;
    * Any ECG finding that, in the opinion of the Investigator, may compromise interpretation of ECG for cardiac safety assessments and/or complicate interpretation of events that may occur post dose (e.g., QT not accurately measurable, conduction abnormalities);
    * QTcF > 470 ms;
    * Any of the following: History or current evidence of congenital long QT syndrome; history of Torsades de Pointes, concomitant medications known to prolong QT interval or history of medication-related QT prolongation;
    * Resting HR <50 bpm or >90 bpm when vital signs are measured at Screening or Admission.
11. COVID-19 positive for active disease.
12. Myocardial impairment of any cause (e.g., cardiomyopathy, ischemic heart disease, significant valvular dysfunction, hypertensive heart disease or congestive heart failure) resulting in heart failure by New York Heart Association (NYHA) Criteria (Class III or IV staging).
13. Current treatment with drugs known as sensitive substrates or substrates having a narrow therapeutic index of CYP2B6, CYP3A4, and transporters including OAT1 and OAT3.
14. Have received inhibitors or inducers of P-gp within 2 weeks prior to receiving the first dose of study drug.
15. Current treatment with drugs which can prolong QTc in adverse reaction.
16. Current treatment with highly competitive protein binding medications, such as warfarin, phenytoin, chlorpromazine, doxorubicin, gentamicin, indomethacin, metoprolol, meclezine.
17. Known hypersensitivity to study drug(s) or any of its constituents.
18. Unwilling or unable to follow study restrictions and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
PART 1: Safety and Tolerability | 12 months
  To characterize the safety and tolerability of DAT-1604 monotherapy by evaluating the number of participants with dose limiting toxicities, adverse events, and laboratory abnormalities as graded by NCI CTCAE version 5.0
PART 2: RP2D | 12 months
  Recommended Phase 2 dose(RP2D) will be definite by safety monitoring committee(SMC).

SECONDARY OUTCOMES:
ORR | 6 months
  Objective Response Rate (ORR) is defined as the proportion of patients that respond either partially or fully to therapy according to RECIST 1.1 criteria based on the CT-Scan.
DCR | 6 months
  Disease control rate (DCR) is defined as the percentage of patients who have achieved CR, PR, Non-CR/Non- PD, or SD in the study.
DOR | 1 year
  Duration of Response (DOR) is defined as the time from the earliest date of documented CR or PR until documented disease progression or death (by any cause, in the absence of progression) as determined by the Investigators using RECIST 1.1.
PFS | 2 years
  Progression-free survival (PFS) is defined as the time from the date of first dose of study drug to the first observation of documented disease progression per RECIST 1.1 as determined by the Investigators or death due to any cause, whichever occurs first.
OS | 2 years
  Overall survival (OS) is defined as the time from the date of first dose of study drug to the date of documented death due to any cause.
AUC | 1 year
  To characterize the single dose PK area under the plasma concentration versus time curve (AUC) of DAT-1604 monotherapy.
Tmax | 1 year
  To characterize the single dose PK time to peak drug concentration (Tmax) of DAT-1604 monotherapy.
Cmax | 1 year
  To characterize the single dose PK peak plasma concentration (Cmax) of DAT-1604 monotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hostital,Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The efficacy and Safety data will be shared.